CLINICAL TRIAL: NCT05908084
Title: A Phase 3 Randomized Study to Compare the Efficacy and Safety of the Humacyte Acellular Tissue Engineered Vessel (ATEV) With That of an Autogenous Arteriovenous Fistula (AVF) in Female Patients With End-Stage Renal Disease Requiring Hemodialysis
Brief Title: To Compare the Efficacy and Safety of the ATEV With AVF in Female Patients With End-Stage Renal Disease Requiring Hemodialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLN-PRO-V012
Expanded Access: NCT03631056 (Approved for marketing)
Record Dates: First submitted 2023-04-28; First posted 2023-06-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: hemodialysis (HD); dialysis catheter
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to either the ATEV or the AVF treatment arm.
Who Masked: Outcomes Assessor
Masking Description: The study team at each site, including the surgeon performing the AVF creation or ATEV implantation, the operating room staff, the dispensing pharmacist, and the Principal Investigator will be unblinded to treatment allocation.
  Members of the Data Monitoring Committee and the Clinical Evaluation Committee, as well as members of the CRO staff may be unblinded to treatment assignment to perform their functions.
  All Sponsor staff, with exception of Chief Medical Officer (CMO) and Head of Biometrics will be unblinded to treatment allocation. Humacyte CMO and Head of Biometrics will be blinded to treatment allocation until the time of the prespecified interim analysis, approximately 12 months after the 80th participant is randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATEV treatment arm (Experimental): ATEV will be implanted as an arterio-venous (AV) access into the forearm or upper arm
  Interventions: Biological: Acellular Tissue Engineered Vessel (ATEV)
- AVF treatment arm (Active Comparator): AVF creation procedure (1-stage AVF or 2-stage AVF) as an arterio-venous (AV) access into the forearm or upper arm
  Interventions: Other: AVF

INTERVENTIONS:
Biological: Acellular Tissue Engineered Vessel (ATEV) — ATEV implantation
  Other Names: Human Acellular Vessel (HAV)
  Arms: ATEV treatment arm
Other: AVF — AVF creation procedure
  Arms: AVF treatment arm

SUMMARY:
The goal of this clinical trial is to compare the number of catheter-free days (CFD) and the rate and severity of any dialysis access-related infections between the ATEV and AVF groups over 12 months in patients with end-stage renal disease (ESRD) needing hemodialysis (HD).

Participants will be stratified by location of the vascular access (forearm versus upper arm) and by type of AVF creation procedure planned by the surgeon at randomization (1-stage AVF versus 2-stage AVF). The comparator is an upper extremity arterio-venous fistula (AVF) for HD access surgically created per the institution's Standard of Care (SoC).

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, two-arm, comparative Phase 3 study of female patients with ESRD, who are receiving clinically successful hemodialysis (HD) via a central venous dialysis catheter (DC).

Approximately 150 female patients will be randomized 1:1 to either the ATEV or the AVF treatment arm. Patients will be stratified by location of the vascular access (forearm versus upper arm) and by type of AVF creation procedure planned by the surgeon at randomization (1-stage AVF versus 2-stage AVF).

All patients will be followed through Month 12 regardless of SA patency status. Patients who have a patent SA at Month 12 will then be followed in the Long-Term Extension study for an additional 12 months with evaluation of exploratory long-term endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with ESRD, currently receiving hemodialysis via dialysis catheter and who are candidates for the creation of an AVF (see Inclusion Criterion #4 below) or implantation of an ATEV for HD access.
2. Patients who plan to undergo HD at a dialysis unit of a participating dialysis provider for at least 12 months after SA creation.
3. Patients aged ≥ 18 years at Screening.
4. Suitable anatomy for creation of a forearm or upper arm AVF and for implantation of straight, curved, or looped ATEV in either the forearm or upper arm.

   NOTE: Suitable anatomy will be determined by both physical examination and ultrasound imaging or vessel imaging modality in addition to consideration of all vascular sites available, prior access failure, future access sites and possibilities to preserve patients' future alternate accesses. Vessel mapping is the preferred method to assess the vascular anatomy, and will evaluate the following attributes during Screening:
   * Vein diameter
   * Arterial diameter
   * Presence of arterial calcification
   * Depth of the intended fistula conduit from the surface of the skin
   * Central vein patency
   * Previous vascular access location The ultimate decision of anatomic suitability belongs to the surgeon and/or the investigator.
5. Hemoglobin ≥ 7 g/dL and platelet count ≥ 100,000 /mm3
6. Patients must either:

   1. Be of non-childbearing potential, which is defined as post-menopausal (at least 1 year without menses prior to Screening) or documented surgically sterile (i.e., total hysterectomy or tubal ligation, or complete bilateral oophorectomy) at least 1 month prior to Screening.
   2. Or, if of childbearing potential:

   Must have a negative serum pregnancy test at Screening, and

   Must agree to use at least one form of the following birth control methods for the duration of the study:

   i. Established use of oral, injectable or implanted hormonal methods of contraception.

   ii. Placement of an intrauterine device or intrauterine system at least 5 days prior to Screening.

   iii. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/ gel/ film/ cream/ suppository.
7. Patient or their legal representative can communicate effectively with investigative staff, is competent and willing to give written informed consent, and able to comply with entire study procedures including all scheduled follow-up visits.
8. Life expectancy of at least 1 year confirmed by Charlson Comorbidity Index ≤ 9.

Exclusion Criteria:

1. Male sex at birth.
2. Planned AVF creation by means other than suture or vascular anastomotic clips (e.g., endovascular surgery or other anastomotic creation devices). Venous outflow from study access cannot be located more distally than the venous outflow of any previous failed access in that extremity.
3. Known serious allergy or intolerance to aspirin and alternative antiplatelet therapy.
4. Pregnancy, or women intending to become pregnant during the course of the trial.
5. Treatment with any investigational drug or device within 60 days or 5 half-lives after taking the last dose (whichever is longer) prior to study entry (Day 1) or ongoing participation in a clinical trial of an investigational product.
6. Documented hyper-coagulable state, as defined as either:

   1. Documented hyper-coagulable state, as defined as either: A biochemical diagnosis (e.g., Factor V Leiden, Protein C deficiency, etc.) - OR -
   2. A clinical history of thrombophilia as diagnosed by 2 or more spontaneous intravascular thrombotic events (e.g., deep vein thrombosis (DVT), pulmonary embolism (PE), etc.) within the previous 5 years.
7. Spontaneous or unexplained bleeding diathesis clinically documented within the last 5 years or a biochemical diagnosis (e.g., von Willebrand's disease, etc.).
8. Cancer actively being treated with a cytotoxic agent.
9. Planned or anticipated renal transplant within 6 months after randomization.
10. Any other condition that in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the SA.
11. Previous exposure to ATEV.
12. Any of the following within 8 weeks prior to screening: acute coronary syndrome, stroke or congestive heart failure NYHA Stage IV
13. Employees of Humacyte and employees or relatives of an investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The number of catheter-free days since randomization to Month 12. | 12 months
  To determine the number of days free from indwelling catheter (catheter-free days) since randomization to 365 days (Month 12), or until SA abandonment, whichever occurs first.
The rate of infections related to any HD access. | 12 months
  To determine the rate of infections, related to any HD access over the period from SA creation (Day 1) until 12 months (365 days) after SA placement, without regard to SA abandonment.

SECONDARY OUTCOMES:
The number of catheter-free days since randomization to Month 6. | 6 months
  To determine the number of days free from indwelling catheter (catheter-free days) from randomization to 183 days (Month 6), or until SA abandonment, whichever occurs first.
The number of days of the study access (SA) functional patency | 12 months
  To determine the number of days of Duration of functional patency of the SA over 12 months from randomization.
The rate of the study access (SA) secondary patency | 6 - 12 months
  To determine the rate of the SA secondary patency at 6 and 12 months from randomization.
The number of days from the study access (SA) maturation to abandonment | 12 months
  To determine the number of days from the study access (SA) maturation to abandonment.
The rate of complications related to any HD access after the study access (SA) creation. | 12 months
  To determine the rate of complications related to any HD access during the 12 months after SA creation, without regard to SA abandonment. For the purposes of this endpoint, HD access refers to any surgically created access or device to provide a route for HD after randomization (e.g., SA, new AVF or AVG, or catheter).

OTHER OUTCOMES:
Incidence rate of HD access-related interventions | 12 months
  Incidence rate of HD access-related interventions over the period from randomization until SA abandonment, or a defined timepoint after randomization (e.g., 12 months).
The number of days from randomization to first day of functional dialysis | 12 months
  To determine the number of days from randomization to the first day of functional dialysis using the SA.
Incidence rate of Study Access (SA) abandonment | 12 months
  To determine the incidence rate of SA abandonment.
Health-related quality of life (HRQoL) of patients (a scale from 0 to 45, with higher scores meaning best outcome) | 12 months
  Health-related quality of life (HRQoL) of patients using the PROMIS-10 Questionnaire, a scale from 0 to 45, where the higher scores mean the best outcome.
Vascular Access Questionnaire (VAQ) score (range 0-68 with higher scores mean worst outcome). | 12 months
  Vascular Access Questionnaire (VAQ) Questionnaire.
  The Vascular Access Questionnaire (VAQ) is a patient reported outcome instrument containing 17 items pertaining to the impact of 17 access-related problems. Responses to the questionnaire are summed to produce a total VAQ score (range from 0-68) with higher values indicating more negative views of vascular access.
The incidence rate of aneurysm or pseudoaneurysm | 12 months
  To determine the incidence rate of clinically significant aneurysm or pseudoaneurysm of the SA over the period from SA creation to 12 months.
The incidence rate of adverse events (AEs) | 12 months
  To determine the incidence rate of adverse events (AEs) from SA creation to 12 months.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Honor Health Scottsdale Shea Medical Center, Scottsdale, Arizona
  - El Centro Regional Medical Center, El Centro, California
  - Jacob's Medical Center at UC San Diego Health, La Jolla, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Access Research Institute, Brooksville, Florida
  - University of FL Health Heart and Vascular Hospital, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - American Access Care of Miami, LLC, Miami, Florida
  - USF Health South Tampa, Tampa, Florida
  - Georgia Nephrology, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - IU Health Bloomington Hospital, Bloomington, Indiana
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers University_Medical, Newark, New Jersey
  - St.Joseph's University Medical Center, Paterson, New Jersey
  - Capital Health Medical Center- Hopewell, Pennington, New Jersey
  - New York-Presbyterian Queens_The Lang Center for Research & Education, Flushing, New York
  - Ambulatory Care Pavilion Westchester Medical Center, Valhalla, New York
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - Duke Regional Hospital, Durham, North Carolina
  - Wake Forest University School of Medicine_Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Dell Seton Medical Center at The University of Texas at Austin, Austin, Texas
  - Dr. Ruben Villa__Nephrology, Lubbock, Texas
  - Cataract & Surgery Center Lubbock, Lubbock, Texas
  - San Antonio Vascular and Endovascular Clinic PLLC, San Antonio, Texas
  - The San Antonio Vascular and Endovascular Clinic, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No